CLINICAL TRIAL: NCT00529997
Title: Clinical Study Comparing Dynamic Stabilization of the Lumbar Spine With the Stabilimax NZ® Dynamic Spine Stabilization System to Posterolateral Instrumented Fusion - In Patients With Lumbar Spinal Stenosis
Brief Title: Dynamic Stabilization for Lumbar Spinal Stenosis With Stabilimax NZ® Dynamic Spine Stabilization System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company has ceased operation
Sponsor: Applied Spine Technologies (Industry)
Responsible Party: Michele Lucey - Vice President of Regulatory Affairs and Quality Assurance, Applied Spine Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AST-A-01; NCT00479544 (obsolete NCT alias)
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Lumbar Spine; Lumbar Spinal Stenosis; Spondylolisthesis; Dynamic Stabilization; Motion Preserving; Arthroplasty; Randomized; Investigational; Back Pain; Leg Pain
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis; Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Posterior Dynamic Stabilization with the Stabilimax NZ
  Interventions: Device: Stabilimax NZ® Dynamic Spine Stabilization System
- 2 (Active Comparator): Posteriolateral instrumented fusion
  Interventions: Device: Stabilimax NZ® Dynamic Spine Stabilization System

INTERVENTIONS:
Device: Stabilimax NZ® Dynamic Spine Stabilization System — Surgical Implantation

SUMMARY:
The purpose of this trial is to assess whether the Stabilimax NZ® is at least as safe and effective as the control therapy of fusion in patients receiving decompression surgery for the treatment of clinically symptomatic spinal stenosis at one contiguous vertebral levels from L1-S1. Safety and effectiveness will be assessed by means of primary study endpoints which address improvements in pain and function in the absence of major device related complications.

The study hypothesis criteria for demonstrating safety and efficacy requires scientific evidence that patients classified as satisfying the primary study endpoint post device implantation is at least as good for Stabilimax NZ® recipients as that for patients undergoing fusion with posterior pedicle screw instrumentation at the 24 month followup assessment.

DETAILED DESCRIPTION:
Degenerative spine disease is a normal part of the aging process. This degeneration can sometimes cause significant pain and limit normal movement.

The pain can be from many sources. For patients being enrolled into this study the pain has been diagnosed to be primarily as a result of a condition called spinal stenosis. The current standard of care for the treatment of moderate to severe spinal stenosis is a surgical procedure that relieves the pressure on the spinal cord and nerves is called decompression surgery. The surgeon removes the tissue and bone that are causing the narrowing thus relieving the pinching of the spinal cord and nerve roots. After surgery, the patient may have a spine that is too unstable. In other words the muscles and ligaments around the spine have to work too hard to maintain normal posture and to control movement. For many years those patients with unstable backs have received fusion therapy. Fusion is the development of bone between the vertebra to stabilize the spine and prevent motion. This is done by inserting a bone graft around the vertebra being treated and placing a rigid brace called a fusion device to prevent movement. Eventually bone will form between the vertebra and the spine will become "fused".

In this study we will be conducting research to evaluate a new, investigative medical device that is designed to brace and support the spine just like fusion but without fusing in the patient's spine. Devices that do this are called "motion preserving" or "dynamic stabilizing" spinal devices. The investigational device that is being evaluated in this study is called the Stabilimax NZ® Dynamic Spinal Stabilization System. The Stabilimax NZ® is inserted and fixed to the vertebra by means of pedicle screws in exactly the same way a fusion device is inserted and attached. The only difference is that for the Stabilimax NZ® no bone graft will be placed around or between the vertebra to promote bone growth for fusion. Patients in the study will receive either the Stabilimax NZ® or will receive a fusion procedure. The study is a randomized controlled clinical trial using a 2:1 investigational:control randomization scheme. The study will enroll 480 patients at approximately 20 investigational sites across the United States.

ELIGIBILITY:
INCLUSION CRITERIA:

Radiographic:

* Degenerative spinal stenosis of the lumbar spine, central, lateral recess, or foraminal;
* Evidence of the cal sac and/or cauda equina compression, nerve root impingement, hypertrophic facets with canal encroachment, with or without spondylolisthesis, if present, no more than grade 1

General:

* The greater of the patients right and left VAS leg pain score is ≥ 40 mm on a 100 mm scale;
* Zurich Claudication Questionnaire Symptom Severity score greater than 2 on a scale of 1-5;
* Zurich Claudication Questionnaire Physical Function score greater than or equal to 2 on a scale of 1-4;
* Intermittent neurogenic claudication
* At least six months of non-surgical management.
* Skeletally mature patients at least 21 years of age;
* Willing to provide written consent for participation and a Health Insurance Portability and Accountability Act authorization;
* Willing to undergo all study procedures including physical therapy and adhere to the follow-up schedule; and
* No additional surgical treatment is required outside the investigational or control at the time of surgery.

EXCLUSION CRITERIA:

Initial Screening:

* Prior surgery at any lumbar level including the level being treated except for: Lamino/Foraminotomy, Microdiscectomy, IDET, and Percutaneous Discectomy.
* Prior surgery at any lumbar level within one year of enrollment;
* No more than one prior surgery at any lumbar level;
* Previous acute trauma at the treated level within two years of enrollment;
* Primary and predominate diagnosis of discogenic back pain, e.g. torn disc, herniated disc inflamed or irritated disc, or other disc pathology;
* Symptomatic cervical and/or thoracic neurological compromise;
* Significant peripheral neuropathy or acute denervation secondary to radiculopathy, caused by conditions other than spinal stenosis;
* Other neurological pathology that could confound study results;
* Cauda Equina Syndrome;
* Contraindicated for MRI;
* Morbid obesity (BMI > 40);
* Peripheral vascular disease requiring intervention (≥ 50% stenosis of vessel);
* Active systemic or surgical site infection;
* Any significant medical conditions that would represent a significant increase in surgical risk or interfere with normal healing;
* History of psychosocial disorders that could prevent accurate completion of self reporting assessment scales
* Women who are pregnant, lactating or anticipate becoming pregnant within 24 months post-surgery;
* Insulin dependent diabetes mellitus;
* Immunocompromised such as but not limited to Acquired Immunodeficiency Syndrome , genetic deficiencies of the complement system, Severe Combined Immunodeficiency Disease, Thymic Hypoplasia;
* Receiving immunosuppressive therapy
* Receiving long-term steroid therapy. Autoimmune disease;
* Active hepatitis;
* Malignancy of any type within the last five years;
* Previous known allergy to the materials contained in the Stabilimax NZ™ device including nickel, cobalt, chromium, molybdenum, iron, titanium, or Teflon™;
* Participation in another clinical study within four weeks of enrollment, or;
* Receiving Worker's Compensation or is involved in active litigation relating to his/her spinal condition;
* Patients who are prisoners.

Radiographic:

* Gross instability, defined as greater than 3 mm translational motion on flexion/extension studies;
* Degenerative spondylolisthesis or retrolisthesis higher than grade 1
* Degenerative scoliosis > 10° at any level(s) in lumbar spine
* Lateral listhesis on A-P X Ray
* Spondylolysis at any level in lumbar spine
* Isthmic Spondylolisthesis at any level in lumbar spine
* Spondylolisthesis at more than one lumbar level;
* DEXA score equal to or below -2.5 T;
* Pathological vertebral fracture;
* Metastases to the spinal vertebra; Paget's disease of bone; Osteomalacia; Pars defect or facet fracture;
* Facet arthropathy at the level(s) to be treated is less than grade 2 and greater than grade 3 according to the Fujiwara scale;
* More than moderate disc degeneration defined as: > 66% loss of disc height compared to the normal, superior adjacent level; and/or moderate to Severe Osteophyte formation;
* Congenital lumbar spinal stenosis;
* Estimated interpedicular distance of less than 30 mm.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2007-02; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Decrease in leg pain of 20 mm on a VAS pain scale; Decrease of ≥ .5 on ZCQ for both Symptom Severity and Physical Function; No major device-related complications; and No surgical revision, reoperation, removal, or supplemental fixation at treated level | 2 years

SECONDARY OUTCOMES:
Reduction in OR Time, Blood Loss, Hospital Stay. Improvement in quality of life and return to work. Improvement in the incidence of adverse events. Radiographic evidence of nonfusion. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Guyer, MD, Principal Investigator — Texas Back Institute; David Musante, M.D., Principal Investigator — Triangle Orthopedics Associates; Neel Anand, M.D., Principal Investigator — Cedars Sinai Medical Center Hospital
Locations (19):
- United States (19):
  - Surgical Specialty Hospital, Phoenix, Arizona
  - Cedars Sinai Medical Center Hospital, Los Angeles, California
  - Tri-City Medical Center, Oceanside, California
  - Littleton Adventist Hospital, Littleton, Colorado
  - New Britain General Hospital, New Britain, Connecticut
  - Morton Plant Mease, Clearwater, Florida
  - Largo Medical Center, Largo, Florida
  - University Community Hospital at Carrolwood, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Upstate Medical Center, Syracuse, New York
  - North Carolina Specialty Hospital, Durham, North Carolina
  - Blanchard Valley Hospital, Findlay, Ohio
  - Sacred Heart Medical Center, Eugene, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Presbyterian Plano Center for Diagnostics & Surgery, Plano, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - DePaul Medical Center, Norfolk, Virginia